CLINICAL TRIAL: NCT01616511
Title: Long-Term Follow-Up for the Pathway CH-1 Trial: Sphenopalatine Ganglion Stimulation for the Acute Treatment of Cluster Headache
Brief Title: Pathway CH-1 Long-Term Follow-Up
Status: Completed | Type: Observational
Sponsor: Autonomic Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-005
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Cluster Headache
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pathway CH-1 Subjects

SUMMARY:
The objective of the study is to demonstrate the long-term safety and performance of the ATI Neurostimulation System when used for stimulation of the sphenopalatine ganglion (SPG) in cluster headache subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been implanted with an ATI Neurostimulator as a part of the Pathway CH-1 trial.
* Subject has completed the Pathway CH-1 Open Label Final office visit and remains implanted with an ATI Neurostimulator.
* Subject has the ability to read, comprehend and to reliably record information as required by the Protocol.
* Subject is able to provide written informed consent prior to participation in the study.

Exclusion Criteria:

* Subject has or requires a pacemaker/defibrillator or other implantable device having a sense amplifier that is programmed 'On.'
* Subject is not suitable for the study for any reason in the judgment of the Investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who have been implanted with an ATI Neurostimulator as a part of the Pathway CH-1 trial, who have completed the Pathway CH-1 trial, and who remain implanted with an ATI Neurostimulator.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2012-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Demonstrate the long-term safety and performance of the ATI Neurostimulation System when used for the stimulation of the SPG in CH Subjects. | Long-Term

CONTACTS AND LOCATIONS:
Overall Officials: Jean Schoenen, MD, PhD, Principal Investigator — Citadelle Hospital
Locations (3):
- Headache Research Unit. University Department of Neurology, Citadelle Hospital, Liège, Belgium
- Danish Headache Center & Department of Neurology, Glostrup Hospital, University of Copenhagen, Glostrup, Copenhagen, Denmark, Denmark
- Servicio de Neurologia, Hospital Clinico Universitario, Valencia, Spain, Spain